CLINICAL TRIAL: NCT04573478
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of Atrasentan in Patients With IgA Nephropathy at Risk of Progressive Loss of Renal Function
Brief Title: Atrasentan in Patients With IgA Nephropathy
Acronym: ALIGN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinook Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHK01-01
Record Dates: First submitted 2020-09-12; First posted 2020-10-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: IgA Nephropathy; Immunoglobulin A Nephropathy
Keywords: Kidney Diseases; Kidney Disease, Chronic; Urologic Diseases; Glomerulonephritis; Glomerular Disease; Glomerulonephritis, IGA; Glomerulopathy; Immunoglobulin Disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases; Renal Insufficiency, Chronic; Urologic Diseases; Glomerulonephritis | interventions — Atrasentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atrasentan (Experimental): Double-blind Period: Once daily oral administration of 0.75 mg atrasentan for 132 weeks.
  Open-label Extension Period: Once daily oral administration of 0.75 mg atrasentan for 48 weeks after completion of 132 weeks on atrasentan or placebo.
  Interventions: Drug: Atrasentan
- Placebo (Placebo Comparator): Double-blind Period: Once daily oral administration of placebo for 132 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atrasentan — Film-coated tablet
  Other Names: CHK-01; Atrasentan Hydrochloride; ABT-627
  Arms: Atrasentan
Drug: Placebo — Film-coated tablet
  Arms: Placebo

SUMMARY:
The ALIGN Study is a phase 3, double-blind, placebo-controlled study to compare the efficacy and safety of atrasentan to placebo in patients with IgA nephropathy (IgAN) at risk of progressive loss of renal function.

DETAILED DESCRIPTION:
Approximately 320 patients with biopsy-proven IgAN will be randomized to receive 0.75 mg atrasentan or placebo daily for 132 weeks. Subjects receive a maximally tolerated and stable dose of a RAS (renin-angiotensin system) inhibitor [such as angiotensin converting enzyme inhibitor (ACEi) or angiotensin-receptor antagonist (ARB)] as part of standard of care. An exception will be made for subjects who are unable to tolerate RAS inhibitor therapy.

Additional subjects receiving a stable dose of SGLT2i will be enrolled to the study. Enrollment in this SGLT2i stable stratum will be in accordance with local regulations in regions that prescribe SGLT2i and will be independent of the 320 subjects enrolled for the primary and secondary analyses.

The primary objective of the study is to evaluate the effect of atrasentan versus placebo on proteinuria as measured by UPCR. Secondary and tertiary objectives include evaluating the change in kidney function over time as measured by eGFR, safety and tolerability, as well as quality of life.

Subjects will have assessments of safety and efficacy over 2 ½ years. To facilitate study participation over this time period, where allowed by local regulations, options for remote study visits using telemedicine and home health may be offered.

Subjects who complete treatment through Week 132 and complete the double-blinded portion of the study may be eligible to enroll in the open label extension of the study to receive atrasentan 0.75 mg daily for up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

Double-Blind period:

* Biopsy-proven IgA nephropathy.
* Receiving a maximally tolerated dose of RAS inhibitor therapy (ACEi or ARB) that has been stable for at least 12 weeks. Exceptions from this requirement will be made for subjects who are unable to tolerate RAS inhibitor therapy.
* Total urine protein ≥1 g/day as measured via 24-hour urine collection by central laboratory at Screening.
* eGFR of at least 30 mL/min/1.73 m^2 at Screening based on the CKD-EPI equation.
* Willing and able to provide informed consent and comply with all study requirements.
* SGLT2i Stable Stratum Only - Receiving a stable dose of an SGLT2i (per Investigator choice) in addition to a maximally tolerated and optimized dose of a RAS inhibitor that has been stable for at least 12 weeks prior to Screening.
* All fertile men and WOCBP who engage in heterosexual intercourse must be willing to abide with highly effective forms of contraception, as specified in the protocol, throughout the study and for 1 month afterward. In WOCBP, use of contraceptive agents must have been started at least 1 month prior to Baseline.

Open-Label Period:

* Willing and able to provide informed consent and comply with all OL extension study visits and study procedures.
* Completed treatment through Week 132 and completed the Week 136 visit.
* All fertile men and WOCBP who engage in heterosexual intercourse must be willing to abide with highly effective forms of contraception, as specified in the protocol, throughout the study and for 1 month afterward. In WOCBP, use of contraceptive agents must have been continued after completing the double-blind portion of the study.

Exclusion Criteria:

Double-blind period:

* Concurrent diagnosis of another cause of chronic kidney disease including diabetic kidney disease or another primary glomerulopathy.
* Clinical diagnosis of nephrotic syndrome.
* BNP value of > 200 pg/mL at Screening.
* Platelet count <80,000 per μL at Screening.
* History of organ transplantation (subjects with history of corneal transplant are not excluded).
* Use of systemic immunosuppressant medications.
* Hemoglobin below 9 g/dL at Screening or prior history of blood transfusion for anemia within 3 months of Screening.

Open-label period:

* eGFR < 25 mL/min/1.73m^2 or evidence of rapidly decreasing eGFR, including unrecovered acute kidney injury or expected to require renal replacement therapy within 3 months
* BNP value of > 200 pg/mL at OL Screening.
* Platelet count < 80,000 per μL at OL Screening.
* Hemoglobin below 9 g/dL at OL screening or prior history of blood transfusion for anemia within 3 months of OL Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Double-blind period: Change in proteinuria | Up to Week 36 or approximately 9 months
  The change in urine protein:creatinine ratio (UPCR) from baseline to Week 36. (non-SGLT2i stratum)
Open-label period: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) | From open-label baseline up to end of treatment visit, 48 weeks
  Type, incidence, severity, seriousness, and relatedness of TEAEs.
Open-label period: Number of Subjects With Adverse Events of Special Interest (AESI) Including Events of Fluid Overload | From open-label baseline up to end of treatment visit, 48 weeks
  Incidence, severity, seriousness, and relatedness AESIs.

SECONDARY OUTCOMES:
Double-blind period: Change in eGFR | Up to Week 136, 4 weeks post end of treatment
  Change from Baseline to final study visit (Week 136, 4 weeks post end of treatment) using the chronic kidney disease-epidemiology collaboration (CKD-EPI) creatinine equation (non-SGLT2i stratum)
Double-blind period: Percent of subjects meeting the first composite endpoint | Up to approximately 2.6 years
  Percent of subjects in the non-SGLT2i stratum meeting the composite endpoint of experiencing at least one of the following during the study:
  * At least a 30% reduction in eGFR sustained for at least 30 days
  * eGFR <15 mL/min/1.73m^2, sustained for at least 30 days
  * Chronic dialysis ≥30 days
  * Kidney transplantation
  * All-cause mortality
Double-blind period: Percent of subjects meeting the second composite endpoint | Up to approximately 2.6 years
  Percent of subjects in the non-SGLT2i stratum meeting the composite endpoint of experiencing at least one of the following during the study:
  * At least a 40% reduction in eGFR sustained for at least 30 days
  * eGFR <15 mL/min/1.73m^2, sustained for at least 30 days
  * Chronic dialysis ≥30 days
  * Kidney transplantation
  * All-cause mortality
Double-blind period: Percent of subjects achieving reduction of proteinuria to < 1 g/day at Week 36 | Baseline to Week 36
  Percentage of subjects with reduction of proteinuria to < 1 g/day and a 25% decrease in total urine protein from Baseline (non-SGLT2i stratum).
Double-blind period: Number of Subjects With TEAEs | From first dose of study drug up to 4 weeks post end of treatment in double-blind period, 136 weeks
  Type, incidence, severity, seriousness, and relatedness of TEAEs.
Double-blind period: Number of Subjects With AESI Including Events of Fluid Overload | From first dose of study drug up to 4 weeks post end of treatment in double-blind period, 136 weeks
  Incidence, severity, seriousness, and relatedness AESIs.
Open-label period: Change in proteinuria | Open-label Baseline to open-label Week 36
  Change in UPCR based on 24-hour urine collection.
Open-label period: Change in eGFR | Open-label Baseline to open-label Week 52
  Change from open-label Baseline to open-label Week 52 using the CKD-EPI creatinine equation.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (135):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Comprehensive Research Institute, Alhambra, California
  - Kidney Disease Medical Group, Glendale, California
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - GA Nephrology Associates, Lawrenceville, Georgia
  - NANI Research, LLC, Hinsdale, Illinois
  - NANI Research, LLC, Fort Wayne, Indiana
  - University of Louisville Physicians- Kidney Disease Program, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Intermed Consultants, Minneapolis, Minnesota
  - Pelican Point Dialysis - DaVita Clinical Research, Las Vegas, Nevada
  - Capital District Renal Physicians, Clifton Park, New York
  - Mountain Kidney and Hypertension Associates, Asheville, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Lehigh Valley Hospital, Bethlehem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Liberty Research Center, Dallas, Texas
  - El Paso Kidney Specialists, El Paso, Texas
  - Nephrology Associates Of Northern Virginia, Fairfax, Virginia
  - Swedish Health Services, Seattle, Washington
- Argentina (4):
  - Centro Médico Ce.Re.Ca, San Luis, San Luis Province
  - CEMIC, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Clinica de Nefrologia Urologia y Enf. Cardiovasculares, Santa Fe
- Australia (8):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Melbourne Renal Research Group, Reservoir, Victoria
  - Sunshine Hospital, Saint Albans, Victoria
  - Box Hill Hospital, Box Hill
  - Royal Brisbane & Women's Hospital, Brisbane
  - Monash Medical Centre, Clayton
  - Renal Research, Gosford
  - Nepean Hospital, Kingswood
- Brazil (7):
  - Instituto Pró-Renal Brasil, Curitiba, Paraná
  - Hospital das Clínicas Universidade Federal de Minas Gerais - UFMG, Belo Horizonte
  - Centro de Pesquisa Clinica do Brasil, Brasília
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Praxis Pesquisa Médica, Santo André
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo
  - Hospital do Rim Fundacao Oswaldo Ramos, São Paulo
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Stephen S. Chow Medicine Professionals, Toronto, Ontario
- China (19):
  - Dongguan Tungwah Hospital, Dongguan, Dongguan
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First A ffliated Hospital of Baotou Medical College, Inner Mangolia University of Science and Technology, Baotou, Inner Mongolia Autonomou
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - People's Hospital of Sichuan Province, Chengdu, Sichuan
  - The First Affiliated Hospital Xinjiang Medical University, Ürümqi, Xinjiang Uygur
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - The Third Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - The Second Hospital of Anhui Medical University, Hefei
  - Shandong University - Qilu Hospital, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Peking University Shenzhen Hospital, Shenzhen
- Colombia (2):
  - Hospital Alma Mater de Antioquia, Medellín, Antioquia
  - IPS Medicos Internistas de Caldas S.A.S, Manizales, Caldas Department
- France (5):
  - CHU de Grenoble - Hopital Albert Michallon, Grenoble
  - CH Emile Roux, Le Puy-en-Velay
  - Hopital Necker, Paris
  - CHU Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Centre Hospitalier Valenciennes, Valenciennes
- Germany (6):
  - St. Josefs-Hospital, Cloppenburg
  - Medizinische Hochschule Hannover, Hanover
  - Nephrologisches Zentrum Hoyerswerda, Hoyerswerda
  - Universitaetsklinikum Jena, Jena
  - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hong Kong (4):
  - Princess Margaret Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong
  - Yan Chai Hospital, Hong Kong
  - The Chinese University of Hong Kong, Shatin
- India (6):
  - Government Medical College, Kozhikode, Kerala
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Christian Medical College, Vellore, Tamil Nadu
  - Osmania General Hospital, Hyderabad, Telangana
  - Yashoda Hospital, Secunderabad, Telangana
  - Nil Ratan Sircar Medical College & Hospital, Kolkata, West Bengal
- Italy (4):
  - Fondazione IRCCS CA Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Seconda Università degli Studi di Napoli, Naples
  - ICS Maugeri SpA SB, Pavia
- Japan (13):
  - Kokura Memorial Hospital (Kokura Kinen Hospital), Fukuoka
  - Kanazawa University Hospital, Kanazawa
  - Nara University, Kashihara
  - St. Marianna University (SMU) School of Medicine, Kawasaki
  - Niigata University, Niigata
  - Okayama University Hospital, Okayama
  - Osaka General Medical Center, Osaka
  - Dokkyo Medical University - Saitama Medical Center, Saitama
  - Showa University Hospital, Shinagawa-ku
  - Juntendo Nerima Hospital, Tokyo
  - Juntendo University Hospital, Tokyo, Tokyo
  - Fujita Health University Hospital, Toyoake
  - Juntendo University Urayasu Hospital, Urayasu
- New Zealand (2):
  - Waikato Hospital, Hamilton
  - Middlemore Clinical Trials, Papatoetoe
- Poland (3):
  - Samodzielny Publiczny ZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego, Lodz
  - Centrum Medyczne Medyk - Rzeszow, Rzeszów
  - Miedzyleski Szpital Specjalistyczny, Warsaw
- Portugal (2):
  - Centro Hospitalar de Lisboa Ocidental EPE - Hospital Santa Cruz, Carnaxide
  - Centro Hospitalar do Medio Tejo (CHMT), E.P.E., Torres Novas
- South Korea (9):
  - Hallym University Medical Center, Anyang
  - Chungnam National University Hospital, Daejeon
  - Myongji Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Jeju National University Hospital, Jeju City
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Severance Hospital, Yonsei University Hospital, Seoul
- Spain (6):
  - Fundacion Puigvert, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital de Sagunto, Sagunto
  - Hospital Universitario Virgen Macarena, Seville
  - H U Dr. Peset, Valencia
- Taiwan (5):
  - Changhua Christian Medical Foundation, Changhua
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University, New Taipei City
  - National Taiwan University Hospital, Taipei
- United Kingdom (7):
  - North Bristol HNS Trust, Clinical Research Centre, Bristol
  - Lister Hospital, Hertford
  - Leicester General Hospital, Leicester
  - King's College Hospital, London
  - Guys Hospital, London
  - Royal London Hospital, London
  - Salford Royal, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heerspink HJL, Jardine M, Kohan DE, Lafayette RA, Levin A, Liew A, Zhang H, Lodha A, Gray T, Wang Y, Renfurm R, Barratt J; ALIGN Study Investigators. Atrasentan in Patients with IgA Nephropathy. N Engl J Med. 2025 Feb 6;392(6):544-554. doi: 10.1056/NEJMoa2409415. Epub 2024 Oct 25. PMID 39460694